CLINICAL TRIAL: NCT00282464
Title: A Six-Week, Double-Blind, Multicenter, Placebo-Controlled Study Evaluating the Efficacy and Safety of Flexible Doses of Oral Ziprasidone in Outpatients With Bipolar I Depression
Brief Title: A Six-week Flexible Dose Study Evaluating the Efficacy and Safety of Geodon in Patients With Bipolar I Depression.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281139
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ziprasidone 20 and 60mg (Active Comparator): For the Ziprasidone arm, the Baseline card will contain 20 mg bid (one 20 mg capsule) for days 1-2 and 40 mg bid (two 20 mg capsules) for days 3-6. Cards A, B, C, and D will contain either 20 mg bid (one 20 mg capsule), 40 mg bid (two 20 mg capsules), 60 mg bid (one 60 mg capsule), or 80 mg bid (one 60 mg capsule and one 20 mg capsule).
  Interventions: Drug: Geodon (Ziprasidone)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Subjects will start on placebo and remain on placebo for six weeks. All cards for the Placebo arm will be 0 mg bid.
  Arms: Placebo
Drug: Geodon (Ziprasidone) — Ziprasidone flexible dosing treatment arm (20-80 mg bid). For the Ziprasidone arm, the Baseline card will contain 20 mg bid (one 20 mg capsule) for days 1-2 and 40 mg bid (two 20 mg capsules) for days 3-6. Cards A, B, C, and D will contain either 20 mg bid (one 20 mg capsule), 40 mg bid (two 20 mg capsules), 60 mg bid (one 60 mg capsule), or 80 mg bid (one 60 mg capsule and one 20 mg capsule).
  Arms: Ziprasidone 20 and 60mg

SUMMARY:
This is a 6-week trial that evaluates the efficacy and safety of Geodon (ziprasidone) in outpatient subjects ages 18 and older with Bipolar Disorder type I, depressed. Subjects are required to undergo a washout period of at least 7 days of any prior med.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a primary diagnosis of Bipolar I Disorder, most recent episode depressed, with or without rapid cycling, without psychotic features, as defined in DSM-IV-TR (296.5X) and confirmed by a structured Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Subjects with a DSM-IV TR diagnosis of schizophrenia (295.XX), schizoaffective disorder (295.70), schizophreniform disorder (295.40), delusional disorder (297.1), or psychotic disorder NOS (298.9).
* Subjects with other DSM-IV TR Axis I or Axis II disorder (in addition to Bipolar I disorder) are ineligible if the comorbid condition is clinically unstable, requires treatment, or has been a primary focus of treatment within the 6 month period prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (42):
  - Pfizer Investigational Site, Dothan, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Darien, Connecticut
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Bradenton, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Eagle, Idaho
  - Pfizer Investigational Site, Granite City, Illinois
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Glen Burnie, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Scranton, Pennsylvania
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia

REFERENCES:
- [Derived] Gao K, Pappadopulos E, Karayal ON, Kolluri S, Calabrese JR. Risk for adverse events and discontinuation due to adverse events of ziprasidone monotherapy relative to placebo in the acute treatment of bipolar depression, mania, and schizophrenia. J Clin Psychopharmacol. 2013 Jun;33(3):425-31. doi: 10.1097/JCP.0b013e3182917f3f. PMID 23609405
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281139&StudyName=A%20six-week%20flexible%20dose%20study%20evaluating%20the%20efficacy%20and%20safety%20of%20Geodon%20in%20patients%20with%20bipolar%20I%20depression.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 day washout: psychotropic drugs and lithium. 4 week washout: monoamine oxidase inhibitors. Depot neuroleptic DC'd 6 months before study entry.11 subjects assigned to but not treated with drug: 9 lost to follow up, 1 no longer willing to participate, 1 DC'd due to protocol violation
Groups:
- Ziprasidone 20-80mg Bid: For the Ziprasidone arm, the Baseline card will contain 20 milligrams (mg) twice daily (bid) (one 20 mg capsule) for days 1-2 and 40 mg bid (two 20 mg capsules) for days 3-6. Cards A, B, C, and D will contain either 20 mg bid (one 20 mg capsule), 40 mg bid (two 20 mg capsules), 60 mg bid (one 60 mg capsule), or 80 mg bid (one 60 mg capsule and one 20 mg capsule).
Period: Overall Study
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Started | 185 | 196
Completed | 112 | 134
Not Completed | 73 | 62
Not completed — Adverse Event | 26 | 20
Not completed — Lack of Efficacy | 8 | 8
Not completed — Lost to Follow-up | 10 | 10
Not completed — Withdrawal by Subject | 24 | 10
Not completed — laboratory abnormality | 1 | 2
Not completed — Protocol Violation | 0 | 7
Not completed — Patient moved | 1 | 0
Not completed — patient non-compliant | 3 | 0
Not completed — patient no show | 0 | 1
Not completed — patient incarcerated | 0 | 1
Not completed — family crisis | 0 | 1
Not completed — dispensed wrong kit | 0 | 1
Not completed — dropped due to missed visits | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone 20-80mg Bid | Placebo | Total
Number analyzed (Participants) | 185 | 196 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.5) | 40.0 (11.7) | 40.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 111 | 219
  Male | 77 | 85 | 162

OUTCOME MEASURES:

1. Secondary Outcome: Response Greater Than or Equal to 50 Percent Decrease From Baseline in Montgomery-Asberg Rating Scale (MADRS) Total Score
Description: Participants with MADRS Total Score greater than or equal to 50 percent decrease from baseline responded yes; others responded no. MADRS: 10-item instrument measuring depression; scale 0(Normal) & 6 (most abnormal)for each item. Total possible score is 0 - 60. Endpoint is last observation carried forward (LOCF)
Time Frame: Baseline to Week 6
Population: Weeks 1 - 6 are Intent to treat (ITT) population Observed Cases
  Not all subjects responded at each week.
  Endpoint is ITT population Last Observation Carried Forward (LOCF)
Measure: Number; unit: participants
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
participants
  Week 1: Yes | 40 | 24
  Week 1: No | 137 | 168
  Week 2: Yes | 55 | 48
  Week 2: No | 105 | 128
  Week 3: Yes | 71 | 60
  Week 3: No | 78 | 105
  Week 4: Yes | 76 | 66
  Week 4: No | 59 | 87
  Week 5: Yes | 81 | 77
  Week 5: No | 40 | 69
  Week 6: Yes | 76 | 83
  Week 6: No | 40 | 58
  Endpoint: Yes | 95 | 97
  Endpoint: No | 85 | 93
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 1; Test type: Superiority or Other; p = 0.0056, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; CMH test stratified by study center and rapid cycling strata was used to compare remission and response rates between ziprasidone and placebo groups
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 2; Test type: Superiority or Other; p = 0.0866, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.0568, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0130, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0188, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.6394, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7707, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Response Greater Than or Equal to 50 Percent Decrease From Baseline in Hamilton Depression Rating Scale (HAM-D 17) Total Score
Description: Participants with greater than or equal to 50 percent decrease from baseline in HAM-D 17 total score responded yes; others responded no. Total score is first 17 items of the HAM-D 25: measures range of depressive symptoms. Scale: 8 items 0-2 & 9 items 0-4, higher scores being more severe. Total possible score is 0 - 52. Endpoint is LOCF.
Time Frame: Baseline to Week 3, Week 6
Population: Weeks 3, 6 are Intent to treat (ITT) population Observed Cases.
  Not all subjects responded at each week.
  Endpoint is ITT population Last Observation Carried Forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
Participants
  Week 3: Yes | 72 | 65
  Week 3: No | 95 | 112
  Week 6: Yes | 85 | 91
  Week 6: No | 41 | 59
  Endpoint: Yes | 95 | 97
  Endpoint: No | 73 | 84
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.2185, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.4124, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6098, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Remission as Measured by Montgomery Asberg Depression Scale (MADRS) Total Score Less Than or Equal to 12
Description: Remission response is yes if MADRS total score less than or equal to 12; if not, response is no. MADRS: 10-item instrument measuring depression; scale 0(Normal) & 6(most abnormal).Total possible score is 0 - 60. Endpoint is LOCF.
Time Frame: Week 1 to Week 6
Population: Weeks 1 - 6 are Intent to treat (ITT) population Observed Cases.
  Not all subjects responded at each week.
  Endpoint is ITT population Last Observation Carried Forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
Participants
  Week 1: Yes | 41 | 21
  Week 1: No | 136 | 168
  Week 2: Yes | 54 | 41
  Week 2: No | 106 | 135
  Week 3: Yes | 70 | 58
  Week 3: No | 79 | 105
  Week 4: Yes | 66 | 60
  Week 4: No | 69 | 93
  Week 5: Yes | 70 | 66
  Week 5: No | 51 | 80
  Week 6: Yes | 70 | 72
  Week 6: No | 46 | 69
  Endpoint: Yes | 87 | 81
  Endpoint: No | 93 | 109
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 1; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 2; Test type: Superiority or Other; p = 0.0099, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.0423, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0618, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0451, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.2633, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.2206, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Remission as Measured by Hamilton Asberg Depression Rating Scale (HAM-D 17) Total Score Less Than or Equal to 7
Description: Remission response is yes when HAM-D 17 total score is less than or equal to 7; if not, response is no. Total score is first 17 items of HAM-D 25, measures range of depressive symptoms. Scale: 8 items 0-2 and 9 items 0-4, higher scores more severe. Total possible score is 0 - 52. Endpoint is LOCF.
Time Frame: Week 3, Week 6
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
Participants
  Week 3: Yes | 32 | 33
  Week 3: No | 135 | 144
  Week 6: Yes | 56 | 51
  Week 6: No | 70 | 99
  Endpoint: Yes | 59 | 55
  Endpoint: No | 109 | 126
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.9863, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.1017, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4033, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: Change is observed value at each visit minus baseline value. MADRS:10-item instrument measuring depression; scale range between 0(Normal) - 6(most abnormal)for each item. Total possible score is 0 - 60. Overall is average response Week 1 - Week 6.
Time Frame: Baseline to Week 6
Population: Weeks 1 - 6 are Intent to treat (ITT) population Observed Cases.
  Overall is Average of Weeks 1 - 6.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 1 (n= 177, 189) | -7.23 (0.79) | -5.02 (0.71)
  Week 2 (n=160, 176) | -9.99 (0.79) | -8.13 (0.72)
  Week 3 (n=149, 163) | -11.88 (0.83) | -10.04 (0.83)
  Week 4 (n=135, 153) | -13.29 (0.92) | -11.53 (0.85)
  Week 5 (n=121, 146) | -14.53 (0.95) | -12.55 (0.88)
  Week 6 (n=116, 141) | -14.88 (1.02) | -13.24 (0.92)
  Overall (n= 180, 190) | -11.97 (0.77) | -10.09 (0.70)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 1; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — No multiple comparison adjustment is applicable. Statistical significance level was 0.05; Fixed categorical: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction & fixed continuous effect of baseline value
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 2; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 4; Test type: Superiority or Other; p = 0.069, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 5; Test type: Superiority or Other; p = 0.053, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6 An estimated sample size of 180 was needed per treatment arm in order to achieve 85% power to detect a treatment difference of 3.5 in the mean change from baseline to Week 6 in MADRS total score with a two-sided t-test at the 0.05 significance level. The common standard deviation was estimated as 11.0. The null hypotheses is equality of mean change from baseline to Week 6 in MADRS total score between ziprasidone and placebo groups; Test type: Superiority or Other; p = 0.154, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Overall; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Change in Hamilton Depression Rating Scale (HAM-D 17) Total Score
Description: Change is observed value at each visit minus baseline value. HAM-D 17 Total score is first 17 items of HAM-D 25; measures range of depressive symptoms patient currently experiencing. Scale: 8 items 0-2 & 9 items 0-4; 0=absent or not depressed, 2 or 4=most severe or extreme. Total possible score is 0 - 52.Endpoint is LOCF
Time Frame: Baseline to Weeks 3, 6
Population: Weeks 3, 6 are Intent to Treat (ITT) population Observed Cases.
  Endpoint is ITT population Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 3 (n=167, 177) | -9.91 (0.88) | -8.73 (0.84)
  Week 6 (n=126, 150) | -12.91 (1.15) | -12.07 (1.06)
  Endpoint (n=168, 181) | -6.92 (1.36) | -7.11 (1.30)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.112, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; ANCOVA model included effects of treatment, rapid cycling, center, prior hospitalization status, as well as baseline value as a covariate
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.352, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.873, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]

7. Secondary Outcome: Change in Total Score in Hamiliton Depression Rating Scale (HAM-D 25)
Description: Change is observed value at each visit minus baseline value. HAM-D: 25-item instrument measuring the range of depressive symptoms patient currently experiencing. Scale: 14 items 0-2 & 11 items 0-4; 0=absent or not depressed, 2 or 4=most severe or extreme. Total possible score is 0 - 72. Endpoint is LOCF.
Time Frame: Baseline to Weeks 3, 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 3 (n=167, 177) | -11.68 (1.07) | -10.76 (1.02)
  Week 6 (n=126, 150) | -15.48 (1.32) | -14.80 (1.22)
  Endpoint (n=168, 181) | -8.06 (1.64) | -8.58 (1.56)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.305, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.510, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.710, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]

8. Secondary Outcome: Change in Bech Melancholia Score
Description: Change is observed value at each visit minus baseline value. Bech Melancholia is sum of scores on 6 Items pertaining to melancholia within HAM-D. Scale range 0 to 4; higher scores, greater severity. Total possible score is 0 - 24. Endpoint is LOCF.
Time Frame: Baseline to Weeks 3, 6
Population: Weeks 3, 6 are Intent to Treat(ITT) population Observed Cases.
  Endpoint is ITT population Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 3 (n =167, 177) | -5.22 (0.50) | -4.28 (0.48)
  Week 6 (n =126, 150) | -6.82 (0.65) | -6.20 (0.6)
  Endpoint (n =168, 181) | -3.73 (0.75) | -3.61 (0.71)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.026, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.223, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.848, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]

9. Secondary Outcome: Change in Anxiety/Somatizations Factor Total Score
Description: Change is observed value at each visit minus baseline value. This test is sum of Scores on 6 Items pertaining to anxiety/somatization within HAM-D. Scale range 0 to 4 with higher scores reflecting greater severity. Total possible score is 0 - 24. Endpoint is LOCF.
Time Frame: Baseline to Weeks 3, 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 3 (n =167, 177) | -2.84 (0.31) | -2.61 (0.30)
  Week 6 (n =126, 150) | -4.09 (0.37) | -3.96 (0.35)
  Endpoint (n =168, 181) | -2.18 (0.43) | -2.57 (0.41)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.381, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.676, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.295, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]

10. Secondary Outcome: Change in Retardation Factor Scores
Description: Change is observed value at each visit minus baseline value. Retardation Factor is the sum of scores of 4 items which pertain to retardation within HAM-D. Scores 0 to 4, higher scores reflecting greater severity.Total possible score is 0 - 16. Endpoint is LOCF.
Time Frame: Baseline to Weeks 3, 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 3 (n =167, 177) | -3.22 (0.35) | -2.68 (0.34)
  Week 6 (n =126, 150) | -4.38 (0.45) | -3.66 (0.42)
  Endpoint (n =168, 181) | -2.24 (0.50) | -1.88 (0.48)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.068, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.043, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.404, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 6, analysis 1]

11. Secondary Outcome: Change in Sleep Disturbance Factor Score
Description: Change is observed value at each visit minus baseline value. Sleep Disturbance is the sum of scores of 3 items which pertain to sleep disturbance within Hamilton Depression Rating Scale (HAM-D). Scale range 0 to 4 with higher scores reflecting greater severity. Total possible score is 0 - 12.
Time Frame: Baseline to Weeks 3, 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 3 (n =167, 177) | -1.51 (0.24) | -1.48 (0.23)
  Week 6 (n =126, 150) | -2.38 (0.28) | -2.31 (0.26)
  Endpoint (n=168, 181) | -1.19 (0.30) | -1.26 (0.29)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.899, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.739, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.797, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]

12. Secondary Outcome: Change in Hamilton Anxiety Rating (HAM-A)
Description: Change is observed value at each visit minus baseline value. HAM-A:14-item scale to rate the intensity of psychic anxiety (items 1- 6, 14) and somatic anxiety (items 7-13) on a 5-point severity scale (0=not present to 4=very severe). Total possible score is 0 - 56.
Time Frame: Baseline to Weeks 3, 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 3 (n=167, 177) | -4.63 (0.69) | -4.18 (0.66)
  Week 6 (n=126, 150) | -6.84 (0.91) | -6.64 (0.84)
  Endpoint (n=168, 181) | -3.05 (1.06) | -3.26 (1.01)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.434, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.777, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.820, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]

13. Secondary Outcome: Change in Total Score of Young Mania Rating Scale (YMRS)
Description: Change is observed value at each visit minus baseline value. YMRS: 11 item instrument with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal; 4 or 8=most abnormal. Total possible score is 0 - 60. Overall is average response Week 1 - 6.
Time Frame: Baseline to week 6
Population: Week 1 - Week 6 is Intent to treat (ITT) population Observed Cases.
  Overall is Average of Weeks 1 - 6.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 1 (n=177, 189) | 0.40 (0.36) | 0.69 (0.33)
  Week 2 (n=160, 176) | 0.49 (0.39) | -0.13 (0.31)
  Week 3 (n=149, 163) | -0.13 (0.41) | 0.00 (0.34)
  Week 4 (n=135, 153) | -0.60 (0.36) | -0.77 (0.31)
  Week 5 (n=121, 146) | -0.94 (0.35) | -0.77 (0.31)
  Week 6 (n=116, 141) | -0.45 (0.43) | -0.66 (0.37)
  Overall (n=180, 190) | -0.20 (0.32) | -0.27 (0.26)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 1; Test type: Superiority or Other; p = 0.468, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 2; Test type: Superiority or Other; p = 0.110, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.738, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 4; Test type: Superiority or Other; p = 0.617, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 5; Test type: Superiority or Other; p = 0.642, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.644, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Overall; Test type: Superiority or Other; p = 0.789, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]

14. Secondary Outcome: Change in Global Clinical Severity of Symptoms (CGI-S)
Description: Change is observed value at each visit minus baseline value. CGI-S is an instrument to measure severity of mental illness. Scale range: 0 = not assessed, 1 = normal, 7 = among most extremely ill
Time Frame: Baseline to week 6
Population: Week 1 - Week 6 is Intent to treat (ITT) population Observed Cases.
  Overall is Average of Weeks 1 - 6.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 1 (n=177, 188) | -0.39 (0.08) | -0.25 (0.07)
  Week 2 (n=160, 176) | -0.66 (0.08) | -0.51 (0.08)
  Week 3 (n=149, 163) | -0.88 (0.10) | -0.84 (0.09)
  Week 4 (n=135, 152) | -1.03 (0.11) | -0.98 (0.10)
  Week 5 (n=121, 146) | -1.27 (0.11) | -1.15 (0.10)
  Week 6 (n=116, 140) | -1.34 (0.11) | -1.28 (0.11)
  Overall (n=180, 190) | -0.93 (0.08) | -0.84 (0.08)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 1; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 2; Test type: Superiority or Other; p = 0.088, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.651, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 4; Test type: Superiority or Other; p = 0.665, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 5; Test type: Superiority or Other; p = 0.349, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.685, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Overall; Test type: Superiority or Other; p = 0.257, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 5, analysis 1]

15. Secondary Outcome: Change in Global Clinical Improvement of Symptoms (CGI -I)
Description: Change is observed value at each visit minus baseline value. CGI-I is an instrument for Global assessment of improvement in patient's condition. Scale range:0=not assessed, 1=very much improved, 7=very much worse
Time Frame: Baseline to Week 6
Population: Week 1 - Week 6 is Intent to treat (ITT) population Observed Cases.
  Overall is Average of Weeks 1 - 6.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 180 | 190
score on scale
  Week 1 (n=177, 188) | 3.37 (0.10) | 3.61 (0.10)
  Week 2 (n=160, 176) | 3.09 (0.11) | 3.29 (0.11)
  Week 3 (n=149, 163) | 2.89 (0.12) | 3.04 (0.11)
  Week 4 (n=135, 152) | 2.74 (0.12) | 2.94 (0.11)
  Week 5 (n=121, 146) | 2.61 (0.13) | 2.84 (0.12)
  Week 6 (n=116, 140) | 2.52 (0.13) | 2.64 (0.12)
  Overall (n=180, 190) | 2.87 (0.10) | 3.06 (0.10)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 1; Test type: Superiority or Other; p = 0.0099, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; Fixed categorical effect: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction
Statistical Analysis 2: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 2; Test type: Superiority or Other; p = 0.0654, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; Fixed categorical effect: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction
Statistical Analysis 3: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 3; Test type: Superiority or Other; p = 0.1807, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; Fixed categorical effect: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction
Statistical Analysis 4: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0957, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; Fixed categorical effect: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction
Statistical Analysis 5: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0752, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; Fixed categorical effect: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction
Statistical Analysis 6: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Week 6; Test type: Superiority or Other; p = 0.3964, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; Fixed categorical effect: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction
Statistical Analysis 7: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Overall; Test type: Superiority or Other; p = 0.0287, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; Fixed categorical effect: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction

16. Secondary Outcome: Change in Global Assessment of Functioning (GAF)
Description: Change is observed value at each visit minus baseline value. GAF is an instrument used to assess global psychological, social, & occupational functioning. Scale range: 100 = normal and 0 = greatest abnormality.
Time Frame: Baseline to week 6 (Endpoint)
Population: Endpoint is ITT population Last Observation Carried Forward (LOCF). n = 154, 169; N = 180, 190
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 154 | 169
score on scale | 9.59 (1.52) | 9.53 (1.42)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Change from baseline to endpoint; Test type: Superiority or Other; p = 0.965, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]

17. Secondary Outcome: Change in Quality of Life, Enjoyment, and Satisfaction Scale (Q-LES-Q) Total Score
Description: Change is observed value at each visit minus baseline value. Q-LES-Q: 16- item instrument for a patient's assessment of his/her quality of life. Scale range: overall level of satisfaction 1=very poor to 5=Very good. 1 item (medication)can be left blank. Total possible score 15 - 80.
Time Frame: Baseline to week 6 (endpoint)
Population: Change from baseline to Endpoint. Endpoint is Intent to Treat (ITT) population Last Observation Carried Forward (LOCF). n = 153, 168; N = 180, 190
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 153 | 168
score on scale | 0.06 (0.02) | 0.06 (0.01)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Change from baseline to endpoint; Test type: Superiority or Other; p = 0.860, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]

18. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score
Description: Change is observed value at each visit minus baseline value. SDS is a patient rated measure of disability and impairment in work/school, social life, family life/home responsibilities. Scale range: 0-10 with 0=no disruption,10=extreme disruption. Total possible score is 0 - 30.
Time Frame: Baseline to week 6 (endpoint)
Population: Baseline to Endpoint. Endpoint is ITT population Last Observation Carried Forward (LOCF). n = 149, 162; N = 180, 190
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 149 | 162
score on scale | -3.69 (0.93) | -3.05 (0.91)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Baseline to endpoint; Test type: Superiority or Other; p = 0.428, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]

19. Secondary Outcome: Change in Bipolar Cognition Rating Scale (BPCoRS) Interviewer Global Rating of Subject
Description: Change is observed value at each visit minus baseline value. BPCoRs: Subject interview with 20-items measuring cognitive deficits & degree of affect on functioning. Scale range:0 to 4, higher numbers, greater impairment. Total possible score is 0 - 80. Endpoint=last observation carried forward (LOCF)
Time Frame: Baseline to week 6 (endpoint)
Population: Baseline to Endpoint. Endpoint is Intent to Treat (ITT) population Last Observation Carried Forward (LOCF). n = 141, 164; N = 180, 190
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 141 | 164
score on scale | -0.65 (0.24) | -0.73 (0.22)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Change from baseline to endpoint; Test type: Superiority or Other; p = 0.708, ANOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; ANOVA model included effects of treatment, rapid cycling, center and prior hospitalization status

20. Secondary Outcome: Change in Bipolar Cognition Rating Scale (BPCoRS) Informant Global Rating
Description: Change is observed value at each visit minus baseline value. Informant Global Rating is interview with informant of subject using BPCoRS, a 20-item instrument measuring cognitive deficits & degree of affect on functioning. Scale: 0 to 4, higher numbers = greater impairment. Total possible score is 0 - 80. Endpoint is LOCF.
Time Frame: Baseline to week 6 (endpoint)
Population: Baseline to Endpoint. Endpoint is ITT population Last Observation Carried Forward (LOCF). n = 97, 104; N = 180, 190
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 97 | 104
score on scale | 4.66 (0.21) | 4.68 (0.21)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.898, ANOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 6, analysis 1]

21. Secondary Outcome: Change in Bipolar Cognition Rating Scale (BPCoRS) Global Rating by Interviewer
Description: Change in Rating by interviewer, using BPCoRS, 20-item instrument measuring cognitive deficits and the degree of affect on functioning; 4 point scale with higher numbers reflecting greater impairment.Total possible score is 0 - 80.
Time Frame: Baseline to week 6 (endpoint)
Population: Endpoint is Intent to Treat (ITT) population Last Observation Carried Forward (LOCF). n = 137, 158; N = 180, 190
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 137 | 158
score on scale | 4.72 (0.18) | 4.63 (0.17)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.559, ANOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; ANOVA model included effects of treatment, rapid cycling, center and prior hospitalization status

22. Secondary Outcome: Change in Bipolar Cognition Rating Scale (BPCoRS) Subject Rating at Endpoint
Description: Change is observed value at each visit minus baseline value. Subject Rating: Subject's perceived change in status using a 20-item instrument measuring cognitive deficits and degree of affect on funtioning. Scale 0 to 4, higher numbers reflecting greater impairment. Total possible score is 0 - 80. Endpoint is last observation carried forward.
Time Frame: Baseline to Week 6 (endpoint)
Population: Endpoint is Intent to Treat (ITT) Last Observation Carried Forward (LOCF). n = 140, 162; N = 180, 190
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Number analyzed (Participants) | 140 | 162
score on scale | 4.69 (0.19) | 4.81 (0.17)
Statistical Analysis 1: Comparison: Ziprasidone 20-80mg Bid vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.458, ANOVA — For all secondary efficacy analyses, no multiple adjustments were made; ANVOVA model included effects of treatment, rapid cycling, center and prior hospitalization status

ADVERSE EVENTS:
Arm/Group | Ziprasidone 20-80mg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 3 | 4
Other Adverse Events (participants affected / at risk) | 93 | 73
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Ziprasidone 20-80mg Bid | Placebo
Skin laceration (Injury, poisoning and procedural complications) | 0/185 | 1/196
Bipolar disorder (Psychiatric disorders) | 0/185 | 1/196
Psychotic disorder (Psychiatric disorders) | 0/185 | 1/196
Suicidal ideation (Psychiatric disorders) | 2/185 | 1/196
Suicide attempt (Psychiatric disorders) | 1/185 | 0/196
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Ziprasidone 20-80mg Bid | Placebo
Diarrhoea (Gastrointestinal disorders) | 8/185 | 15/196
Nausea (Gastrointestinal disorders) | 11/185 | 21/196
Fatigue (General disorders) | 13/185 | 8/196
Dizziness (Nervous system disorders) | 12/185 | 10/196
Headache (Nervous system disorders) | 21/185 | 21/196
Sedation (Nervous system disorders) | 22/185 | 6/196
Somnolence (Nervous system disorders) | 25/185 | 5/196
Depression (Psychiatric disorders) | 6/185 | 13/196
Insomnia (Psychiatric disorders) | 9/185 | 10/196

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.